CLINICAL TRIAL: NCT01857336
Title: Infusion of Recombinant Human Granulocyte Colony Stimulating Factor Mobilized Peripheral Harvest for Poor Engraftment After Hematopoietic Stem Cell Transplantation
Brief Title: G-CSF Moblized Peripheral Harvest for Poor Engraftment After Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-03
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Poor Graft Function; Stem Cell Transplantation; Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- infusion group (Experimental): Patients with PGF were planed to infusion peripheral harvest. The peripheral cell harvest was aphaeresis on the fourth or fifth day after mobilization with recombinant human granulocyte colony stimulating factor.
  Interventions: Other: infusion of G-CSF mobilized peripheral harvest

INTERVENTIONS:
Other: infusion of G-CSF mobilized peripheral harvest

SUMMARY:
Poor graft function (PGF) is a common complication after allogeneic stem cell transplantation, which was associated with high mortality. The pathogenesis fo PGF was poorly understood. Infusion of donor peripheral cell harvest was effective for some patients with PGF in our preliminary study. This present study aimed to explore the efficacy of peripheral cell harvest for poor graft function.

DETAILED DESCRIPTION:
Poor graft function (PGF) is a common complication after allogeneic stem cell transplantation, which was associated with high mortality. The pathogenesis fo PGF was poorly understood. Infusion of donor peripheral cell harvest was effective for some patients with PGF in our preliminary study.The peripheral cell harvest was aphaeresis on the fourth or fifth day after mobilization with recombinant human granulocyte colony stimulating factor. Hematogical response was assessed at 30 days after infusion. Good response was defined as neutrophil > 1.0×109/l without G-CSF support for at least 3 consecutive days, and persistent platelet >20×109/l without transfusion for at least 7 days. Otherwise, poor response was defined.

ELIGIBILITY:
Inclusion Criteria:

* patients received allogeneic stem cell transplantation;diagnosis of PGF after HSCT; without concurent GVHD,RELAPSE of underlying disease.

Exclusion Criteria:

* age<14 years;active GVHD;relapse of underlying disease

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
hematological response | 30 days after infusion
  Hematogical response was assessed at 30 days after infusion. Good response was defined as neutrophil > 1.0×109/l without G-CSF support for at least 3 consecutive days, and persistent platelet >20×109/l without transfusion for at least 7 days. Otherwise, poor response was defined.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China